CLINICAL TRIAL: NCT02437565
Title: Checking Occlusion During Stainless Steel Crown Placement in Children Under General Anesthesia - Evaluation of a Novel Technique
Brief Title: Checking Occlusion During Stainless Steel Crown Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr Sharat Pani, Assistant Professor, Pediatric Dentistry, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRP/2013/046
Record Dates: First submitted 2015-04-24; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Placement of stainless steel crown under general anesthesia without the use of an occlusal template
  Interventions: Other: Stainless steel crown
- Impression (Experimental): Placement of stainless steel crown under general anesthesia with the use of an occlusal template prepared after making an impression of the teeth using a fast setting polyvinyl siloxane material
  Interventions: Other: Stainless steel crown; Other: Occlusal Template

INTERVENTIONS:
Other: Stainless steel crown — Placement of stainless steel crowns for teeth that have undergone pulpotomy for the treatment of pulpitis induced by severe early childhood caries under general anesthesia
Other: Occlusal Template — Use of an occlusal template for the placement of stainless steel crowns under general anesthesia
  Arms: Impression

SUMMARY:
Stainless steel crowns are arguably the most successful posterior restorations in primary teeth and have been so for more than 50 years. Stainless steel crowns offer durability and success rates in excess of 95% making them the restoration of choice for posterior primary teeth in children treated under general anesthesia.

Failures of stainless steel crowns placed on primary teeth have been documented using several criteria including marginal adaptation, recurrent caries, abscess formation or root resorption, loss of the crown due to faulty retention and even perforation of the crown . Despite the probability that factors such as root resorption and failure of endodontic treatment could be due to traumatic occlusion, surprisingly little evidence is available in literature on the attempts made to check or evaluate the occlusion of stainless steel crowns placed under general anesthesia The aim of this study was to compare the time taken for placement and the overall success of bilateral multiple stainless crowns placed under general anesthesia using an occlusal index and compare them to crowns placed without such an index, using a randomized control study design

DETAILED DESCRIPTION:
A total of 60 patients (32 male and 28 female) aged between 4 and 7 years (Mean age 4.8 years, SD +/- 1.09 years) who met the inclusion criteria were recruited after obtaining informed consent from the parent. No financial incentives were offered for participation in the study. A total of 51 (29 male and 22 female) patients completed the six month follow up requirement (Fig 2).

Evaluation Crowns and the Procedure All patients were evaluated at 24 hours, one week, three months and six months post-operatively. Clinical criteria evaluated included the reporting of pain, discomfort, difficulty in mastication or high points reported by the patient. Tenderness on percussion, presence of premature mobility and clinical evidence of an abscess or fistula were checked by one of the investigators (SCP). Periapical digital radiographs were taken using a digital sensor (Schick Elite, Sirona Dental Inc. Long Island NY. USA) and were evaluated by the same examiner for radiographic evidence of failure. In order to ensure blinding the investigator (SCP) recording the findings was not made aware of which group the patient belonged to. The time taken for each procedure was calculated from the time of placement of the throat pack to the time of removal of the throat pack and was obtained from the intra-operative anesthesiologist notes. If failure of the crown occurred at 3 months, these teeth were excluded from the 6 month evaluation.

Statistical Analyses The parametric values of the control and case groups were compared using the student's t test. The non-parametric values of the control and case groups were compared using the Mann Whitney U test. All tests were conducted at p value of 0.05

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Severe Early Childhood Caries
* Have behavioral problems that require management under general anesthesia
* ASA class I
* Deep Dental Caries involving the pulp in all eight primary molars

Exclusion Criteria:

* ASA class II or above
* Initial treatment plan cannot be carried out
* Need for extraction or pulpectomy in one or more primary molar

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time taken for the completion of oral rehabilitation | Measured at the end of the clinical procedure
  Time taken for the completion of oral rehabilitation under general anesthesia

SECONDARY OUTCOMES:
Discomfort on Biting | up to 6 months
  Patient complains of discomfort on biting
Radiographic Evidence of Abscess | up to 6 monhts
  Presence of abcess on a periapical radiograph
Dislodgement of crown | up to 6 months
  Loss of retention of the crown resulting in the dislodgement or complete removal of crown

CONTACTS AND LOCATIONS:
Overall Officials: Sharat C Pani, MDS, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia